CLINICAL TRIAL: NCT01590485
Title: Evaluation of the Effect of Saffron (Crocus Sativus) on Pain Control After Root Canal Therapy in Teeth With Vital Pulps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zahedan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Kaveh Oloomi, DDS, MS, Assistant Professor, Zahedan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: pain control by saffron
Record Dates: First submitted 2012-04-27; First posted 2012-05-03 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Post-treatment Pain Following Root Canal Therapy
Keywords: pain; root canal therapy
MeSH Terms: conditions — Pain | interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Starch capsule (Placebo Comparator): starch with dose of 100 mg in each capsule every 6 hours up to 48 hours (400 mg/day)
  Interventions: Other: starch
- Saffron capsule (Active Comparator): saffron with dose of 100 mg in each capsule every 6 hours up to 48 hours (400 mg/day)
  Interventions: Other: saffron

INTERVENTIONS:
Other: starch — 100 mg in each capsule every 6 hours up to 48 hours (400 mg/day)
  Arms: Starch capsule
Other: saffron — 100 mg in each capsule every 6 hours up to 48 hours (400 mg/day)
  Other Names: Crocus sativus
  Arms: Saffron capsule

SUMMARY:
The purpose of this study is to determine whether saffron is effective in the pain control after root canal therapy in vital teeth.

DETAILED DESCRIPTION:
Among patients refer to endodontics department of Zahedan Faculty of Dentistry whom with moderate to severe pain in a single canal tooth will be selected and randomly divided in 2 groups of saffron and placebo. After root canal therapy each patient in each group will receive a box of 8 similar capsules. They will use 1 capsule exactly after treatment completion and then each 6 hours up to 48 hours. Patients will record their pain intensity in each time period according to Visual Analog Scale(VAS)and finally mean pain intensity will be compared between 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* patients who have at least one vital tooth with one root canal and moderate to severe pain

Exclusion Criteria:

1. teeth with periapical lesions
2. patients with history of:

   * allergy to saffron
   * diabetes mellitus
   * cardiovascular disorders
   * kidney and liver diseases
   * blood and hormonal disorders
   * electrolyte imbalance
3. women in pregnancy or breast feeding period and
4. use of analgesics or opioids during 4 hours before treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
change in VAS score | Every 6 hours after treatment completion up to 48 hours
  Patients will record their pain intensity in each time period according to Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Kaveh Oloomi, DDS, MS, Principal Investigator — Zahedan University of Medical Sciences
Locations (1):
- Zahedan university of medical sciences, Vice-chancellor for research, Zahedan, Iran